CLINICAL TRIAL: NCT06906900
Title: A Phase I Study of the NovoTTF-200M and Novo TTF-200A Systems for the Treatment of Refractory Spinal Metastasis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1879; NCI-2025-02319 (Other: NCI-CTRP Clinical Trials Registray)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Spinal Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with 150 KHZ (NovoTTF-200M) or 200KHZ (NovoTTF-200A) (Experimental)
  Interventions: Device: TTF-200M and TTF-200A systems

INTERVENTIONS:
Device: TTF-200M and TTF-200A systems — Participants will receive one cycle and treatment will continue as long as the doctor thinks it is in the participant's best interest.

SUMMARY:
This clinical research study is to learn about the safety of the NovoTTF-200M and Novo TTF-200A Systems, when used either alone or in combination with standard therapy, in patients with tumors that did not respond to treatment.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the safety of applying TTFields at frequencies between 150 and 200KHz, using the TTF200M and TTF-200A systems (respectively), alone or in combination with available systemic therapies as adjuvant treatment in patients with radiation refractory spinal metastasis. Safety will be specifically assessed based on absence of wound dehiscence in the surgical group and severe cellulitis requiring drainage and intravenous antibiotics in both surgical and non-surgical cohorts.

Secondary Objective:

To assess local spine progression-free survivals at about every 3 months (+/- 1 month) in these patients until one of the following occurs: local disease progression, transition to hospice, loss of follow up, withdrawal from study or consent, whichever comes first.

Exploratory Objectives:

1. To evaluate the safety of application of tumor treating fields at frequencies between 150kHZ and 200 KHZ using the TTF-200M and TTF-200A systems (respectively), alone or in combination with available systemic therapy as adjuvant treatment after surgery for spinal cord decompression in patients with refractory spinal metastasis
2. To assess local spine progression-free survivals at about every 3 months (+/- 1 month) until their local disease progresses, they go to hospice, or are off study, whichever is earlier, in patients in 2.3(a).
3. To evaluate the safety of application of tumor treating fields at frequencies between 150kHZ and 200 KHZ using the TTF-200M and TTF-200A systems (respectively), alone or in combination with available systemic therapy as adjuvant treatment for patients with radiation refractory spinal metastasis who are unable to undergo surgery due to high risk of complications.
4. To assess local spine progression-free survivals at about every 3 months (+/- 1 month) until their local disease progresses, they go to hospice, or are off study, whichever is earlier, in patients in 2.3(c).
5. To evaluate change in plasma ctDNA levels before initiation (baseline) to Cycle 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one or more spinal metastasis(es) affecting levels between C1 to S4 which have been previously treated with surgery and/or maximal doses radiation therapy to the spinal metastasis. For patients in the surgical group, patients must have completed maximal intralesional debulking of their tumor (within 90 days of enrollment).
2. No more radiation options available for treatment to the spinal metastasis(es) that will undergo the TTF treatment
3. Male or Female subjects aged ≥ 22 years.
4. Women of child-bearing potential (women who are not postmenopausal for at least one year or are not surgically sterile) must agree prior to study entry to use adequate contraception (e.g., hormonal, barrier device, or abstinence) for the duration of study participation.
5. Patients must have a Karnofsky Performance Scale (KPS) (Appendix D) score of at least 70%.
6. Patients must have the ability to independently disconnect the arrays or turn off the system if they feel uncomfortably hot while using the device.
7. Patients (and/or legally authorized representative) should be able to fully understand the requirements of the trial, including the need to use the device for at least 18 hours per day, be willing to comply with all trial visits and assessments and be willing and able to sign an Institutional Review Board (IRB) approved written informed consent document (or provide assent where applicable).
8. Patients with the following tumor histologies (numbers in parenthesis represent the frequencies/device patients with these histologies will be treated with):

   1. Non-small cell lung cancer (150KHZ, TTF-200M)
   2. Chordoma (150KHZ, TTF-200M)
   3. Breast adenocarcinoma (150HKZ, TTF-200M)
   4. Liver/gastrointestinal malignancy (150 KHZ, TTF-200M)
   5. Endocrine origin carcinoma (150KHZ, TTF-200M)
   6. Renal cell carcinoma (200KHZ, TTF-200A)
   7. Prostate adenocarcinoma (200KHZ, TTF-200A)
   8. Sarcoma (200KHZ, TTF-200A)
9. For the non-surgical group only, expected survival of more than 8 months as confirmed by the primary oncologist.
10. For the non-surgical group only, in case of multiple noncontiguous vertebral levels requiring treatment, all sites must be included under the largest length of the antero-posterior set of transducer arrays (25cm).
11. Patients who have previously undergone surgery and already have spinal hardware implanted in the intended area of treatment may be enrolled in the surgical group, regardless of the timing of their original surgery.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will not be eligible for the study:

1. Psychiatric illness/social situations (homeless or living in a foreign country) that would limit compliance with study requirements.
2. Physical or cognitive limitation that prevents the ability to independently disconnect the arrays or turn off the system if they feel uncomfortably hot while using the device. This includes patients that need a legally authorized representative for consent.
3. Patients in the surgery group who have not fully recovered from the spinal surgery, where wound healing is compromised, requiring healing by second intention (i.e., the wound is left open and heals spontaneously).
4. History of allergic reactions or sensitivity to conductive hydrogels used on electrocardiogram (ECG) stickers or transcutaneous electrical nerve stimulation (TENS) electrodes.
5. Implanted pacemaker, defibrillator, nerve stimulator or other active electronic medical devices in the area of surgery or application of the skin transducers.
6. Women who are pregnant or lactating.
7. Prior surgery to the spinal level(s) to be treated with TTF is not an exclusion criterion.
8. Enrollment on another clinical trial with investigational drugs/devices is not an exclusion criterion and is kept at the discretion of the treating surgeon.
9. Patients with leptomeningeal disease.
10. Patients with severe pre-existing dermatological conditions (i.e., active herpes zoster, bullous pemphigoid reactions, Stevens-Johnson syndrome) that might interfere with interpretation of the device's skin toxicity.
11. Patients receiving targeted therapy (i.e., EGFR inhibitors) who present with severe dermatological reactions at the site(s) to receive treatment with NovoTTF-200A or NovoTTF-200M. Prior treatment and complete resolution of a prior severe dermatological reaction are not exclusion criteria.
12. Multiple noncontiguous progressive spine tumors separated by more than 25 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-02-17 (Estimated); Study Completion 2029-02-17 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Tatsui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org